CLINICAL TRIAL: NCT01846325
Title: The Effects of Administration of Combined Docosahexaenoic Acid and Vitamin E Supplements on Spermatogram and Seminal Plasma Oxidative Stress in Infertile Men With Asthenozoospermia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Dr, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 046401
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Asthenozoospermia
MeSH Terms: conditions — Asthenozoospermia | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- DHA plus vitamin E (Experimental): Cap DHA 460mg plus vitamin E 600mg per day
  Interventions: Dietary Supplement: vitamin E; Dietary Supplement: DHA
- VitaminE plus placebo (Active Comparator): vitamin E 600 mg plus placebo
  Interventions: Dietary Supplement: vitamin E; Other: placebo
- placebo plus placebo (Placebo Comparator): DHA shaped placebo plus vitamin E shaped placebo
  Interventions: Other: placebo
- DHA plus placebo (Active Comparator): 460 mg DHA plus placebo
  Interventions: Dietary Supplement: DHA; Other: placebo

INTERVENTIONS:
Dietary Supplement: vitamin E
  Arms: DHA plus vitamin E; VitaminE plus placebo
Dietary Supplement: DHA
  Arms: DHA plus placebo; DHA plus vitamin E
Other: placebo
  Arms: DHA plus placebo; VitaminE plus placebo; placebo plus placebo

SUMMARY:
Since docosahexaenoic acid (DHA) level in sperm membrane has been shown to be decreased in asthenozoospermic men, the investigators hypothesized that DHA supplementation may improve it. Furthermore, the investigators added vitamin E to it to protect its unsaturated bonds which are susceptible to oxidation and production of free oxygen radicals.

ELIGIBILITY:
Inclusion criteria:

* Willing to participate in the study and filling out the informed consent form
* should be infertile (no conception after 12 months intercourse without any contraception)
* age 20-45 y.o, idiopathic asthenospermia according to WHO criteria
* normal hormonal profile

Exclusion criteria:

* any infection in genitourinary (GU) tract
* any anatomical abnormality in GU tract
* any chronic disease during last 3 months
* any surgery in GU tract
* consumption of omega-3 fatty acids and/or vitamin E supplements during last 3 months

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
sperm motility | 12 weeks
  spermatogram

SECONDARY OUTCOMES:
sperm count | 12 weeks
  spermatogram
seminal oxidative stress | 12 weeks
  ELISA

REFERENCES:
- [Derived] Eslamian G, Amirjannati N, Noori N, Sadeghi MR, Hekmatdoost A. Effects of coadministration of DHA and vitamin E on spermatogram, seminal oxidative stress, and sperm phospholipids in asthenozoospermic men: a randomized controlled trial. Am J Clin Nutr. 2020 Sep 1;112(3):707-719. doi: 10.1093/ajcn/nqaa124. PMID 32453396